| Participant ( | Consent | <b>Form</b> |
|---------------|---------|-------------|
|---------------|---------|-------------|

| Study Number |
|--------------|

Safety and efficacy of low elasticity polyvinylidene fluoride (DynaMesh®-SIS soft) retropubic tension free midurethral sling in the treatment of stress urinary incontinence in women.

| 1. | I confirm that I have read and understand the information sheet dated (version ) for the above study. I have had the |
|---|---|
| | opportunity to consider the information, ask questions and have had these answered satisfactorily. |
| | Initial box |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. |
| | Initial box |
| 3. | I understand that relevant sections of my medical notes and data collected during the study may be looked at by individuals from this hospital, the main research centre and from Kebomed UK. I give permission for these individuals to have access to my records. |
| | Initial box |
| 4. | I agree to my GP being informed of my participation in the study. |
| | Initial box |
| 5. | I agree to my GP being informed if there are any concerns about my physical or mental health raised from my questionnaires or examinations |
| | Initial box |
| 6. | I agree to take part in the above study. |
| | Initial box |
| Nam | ne of participant in full: |
| Date | »: |
| Sign | ature: |
| Nam | ne of person taking consent: |
| Date | »: |
| Sian | ature: |